CLINICAL TRIAL: NCT07243782
Title: Regulatory Post-Marketing Surveillance to Assess Safety and Effectiveness in Hidradenitis Suppurativa, Pediatric Plaque Psoriasis and JIA Treated With Cosentyx®(Secukinumab) in Korea : a rPMS Study
Brief Title: Regulatory Post-Marketing Surveillance in Hidradenitis Suppurativa, Pediatric Plaque Psoriasis and JIA Treated With Cosentyx®(Secukinumab) in Korea
Status: Not yet recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457MKR01
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hidradenitis Suppurativa; Pediatric Plaque Psoriasis; Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Hidradenitis Suppurativa; Arthritis, Juvenile | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Secukinumab - HS: Participants with Hidradenitis Supurativa who are receiving or will receive Cosentyx after the start of this study in routine clinical practice.
  Interventions: Drug: Secukinumab
- Secukinumab - Pediatric plaque psoriasis: Participants with pediatric plaque psoriasis who are receiving or will receive Cosentyx after the start of this study in routine clinical practice.
  Interventions: Drug: Secukinumab
- Secukinumab - JIA: Participants with juvenile idiopathic arthritis who are receiving or will receive Cosentyx after the start of this study in routine clinical practice.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — This is a prospective observational study. There is no treatment allocation. The decision to initiate treatment will be based solely on clinical judgement.
  Other Names: Cosentyx

SUMMARY:
Regulatory Post-Marketing Surveillance in hidradenitis suppurativa, pediatric plaque psoriasis and JIA treated with Cosentyx®(secukinumab) in Korea

DETAILED DESCRIPTION:
This post-marketing study is a multicenter, single-arm, prospective, observational study.

Cosentyx is prescribed within the scope of the approved indications for hidradenitis suppurativa, pediatric plaque psoriasis, enthesitis-related arthritis and juvenile psoriatic arthritis in the juvenile idiopathic arthritis category. The decision to treat patients with the drug will be made within current clinical practice and will be clearly distinguished from the decision to include patients in this investigation. No additional diagnostics or monitoring will be performed for this study beyond what is typically performed in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Hidradenitis suppurativa:

1. Adults 18 years of age and older with moderate to severe hidradenitis suppurativa who are or will be receiving Cosentyx within the scope of approved indication.
2. Patients who have agreed to participate in study (written informed consent)

Pediatric plaque psoriasis:

1. Patients with moderate to severe plaque psoriasis between the ages of 6 and 18 years who are receiving or will receive Cosentyx within the scope of approved indication.
2. Patients with patient or guardian consent to participate in study (written informed consent)

Juvenile idiopathic arthritis:

1. Enthesitis related arthritis and juvenile psoriatic arthritis in juvenile idiopathic arthritis category patients with enthesitis related arthritis and juvenile psoriatic arthritis in juvenile idiopathic arthritis category between the ages of 6 and 18 years and are receiving or will receive Cosentyx within the scope of approved indication.
2. Patients with patient or guardian consent to participate in study (written informed consent)

Exclusion Criteria:

1. Patients who are contraindicated according to national prescribing information
2. Patients participating in other interventional clinical trials

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are receiving or will receive Cosentyx after the start of this study in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants having Adverse Events (AEs) and Serious Adverse Events (SAEs) within each indication | Up to 24 weeks
  All AEs, regardless of severity or causality, will be collected from all participants enrolled in the study.

SECONDARY OUTCOMES:
Proportion of paticipants achieving 50% reduction in hidradenitis suppurativa clinical response (HiSCR50) - HS participants | 12 and 24 weeks
  The HiSCR is a validated assessment tool developed for patients with hidradenitis suppurativa. It is a dichotomized clinical response assessment that measures the status of three types of lesions: abscesses, inflammatory nodules, and draining fistulas. HiSCR50 is defined as participants who have at least a 50% reduction in abscess and nodule count compared to baseline and no increase in the number of abscesses or draining tunnels.
Proportion of participants achieving a severity of 0 or 1 on the hidradenitis supurativa-physician's global assessment (HS-PGA) - HS participants | 12 and 24 weeks
  The HS-PGA is a global assessment of patients with hidradenitis suppurativa based on four clinical assessments [number of abscesses, number of draining fistulas, number of inflammatory nodules, and presence/absence of non-inflammatory nodules] to determine severity on a six-point scale, scores range from 0-5 based on the number of HS lesions ranges from clear to very severe.
Proportion of participants with a 55% or greater reduction in international hidradenitis suppurativa severity scoring system (IHS4-55) - HS participants | 12 and 24 weeks
  The IHS4 is an exclusively physician-based, clinical scoring system for dynamic assessment of HS severity.
  HS severity is calculated based on the number of lesions multiplied by their respective score: the IHS4 score (points) = (number of nodules multiplied by 1) + (number of abscesses multiplied by 2) + [number of draining tunnels (fistulae/sinuses) multiplied by 4].
  HS4-55 is defined as participants who have at least a 55% reduction in IHS4 score compared to baseline.
Proportion of participants with a ≥30% reduction in Hidradenitis suppurativa-related skin pain numerical rating scale (NRS) - HS participants | 12 and 24 weeks
  The HS-related skin pain NRS is a numeric rating scale in which patients rate their pain at the time of the worst skin pain in the past 24 hours. The numeric rating scale is a fine-grained numeric version of a visual analogue scale (VAS) in which respondents select a number (0-10) that best reflects the intensity of their pain, ranging from 0 (no skin pain) to 10 (most severe skin pain)
Proportion of participants with an Hidradenitis supurativa flare - HS participants | 12 and 24 weeks
  An HS flare is a new or substantial worsening of clinical signs or symptoms.
Proportion of participants by Hurley stage - HS participants | 12 and 24 weeks
  The Hurley stage is a grading system for classifying the severity of hidradenitis suppurativa. Stage I is defined as abscess formation (single or multiple), no sinus tracts or cicatrization/scarring, Stage II is defined as recurrent abscesses with sinus tracts and scarring, single or multiple separated lesions, and Stage III is defined as diffuse or almost diffuse involvement, or multiple interconnected sinus tracts and abscesses across the entire area.
Change from baseline in Psoriasis Area and Severity Index (PASI) - Pediatric plaque psoriasis participants | 12 and 24 weeks
  The PASI is a composite index that combines the area of involvement of psoriatic lesions with the severity of the lesions. The PASI calculates the extent of redness/erythema, scaling, and thickness/thickness of psoriatic lesions and assesses their severity with a corresponding score. PASI scores can range from a lower value of 0, corresponding to no signs of psoriasis, up to a theoretic maximum of 72.0.
Proportion of participants achieving an Investigator's Global Assessment (IGA) score of 0 or 1 - Pediatric plaque psoriasis participants | 12 and 24 weeks
  The IGA mod 2011 score is used to determine the severity psoriasis symptoms. It reflects a subject's overall disease severity for the whole body. The scale includes 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe.
Change from baseline in active joints by Tender Joint Count (TJC) - JIA participants | 12 and 24 weeks
  A joint is classified as "active" when there is swelling, pain on movement, tenderness/pain on movement, and limitation of motion. It is also possible to classify a joint as "active" if only edema is present.
  Using digital pressure, joints that feel tender or show pain when moved are considered tender joints, and their counts are totaled to determine the tender joint count (TJC).
Change from baseline in active joints by swollen joint count (SJC)- JIA participants | 12 and 24 weeks
  A joint is classified as "active" when there is swelling, pain on movement, tenderness/pain on movement, and limitation of motion. It is also possible to classify a joint as "active" if only edema is present.
  Swollen joint count SJC is determined by physical examination of joint counts that are classified as either swollen or not swollen.
Change from baseline in clinical juvenile arthritis disease activity score (cJADAS) - JIA participants | 12 and 24 weeks
  The JADAS is a tool for assessing disease activity in Juvenile idiopathic arthritis that is composed of four items: joint count (number of active joints as assessed by a physician), physician global assessment of disease activity (VAS 0-10), parent/patient global assessment (VAS 0-10), and serum inflammatory markers (erythrocyte sedimentation rate (ESR)), which are scored separately and summed to calculate a score. The clinical JADAS (cJADAS) used in this study excludes serum inflammatory markers and is calculated by summing all the scores (0-10) obtained from each item, and the score is calculated from a minimum of 0 to a maximum of 30.
Physician evaluation of participant symptoms | 12 and 24 weeks
  Treatment effect is evaluated by physician based on clinical judgement and/or laboratory test results and classified in four categories.
  * Improved: improvement or maintenance of symptoms*, as determined by the investigator.
  * Unchanged: No significant change from pre-initiation of the investigational drug is identified, which is not considered a maintenance effect*.
  * Worsening: Symptoms are worse than before started taking the investigational drug.
  * Unevaluable: Unable to evaluate due to lost to follow-up, etc. * Maintenance effect: When there is a significant risk of worsening of symptoms if the medication is discontinued, or when substitution with an existing medication continues to have an equivalent effect.

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com